CLINICAL TRIAL: NCT05358197
Title: Investigation of the Effect of Laughter Yoga on Sleep Quality and Happiness in Individuals
Brief Title: Effect of Laughter Yoga on Sleep Quality and Happiness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Kevser Sevgi Ünal Aslan, Nursing Department, Osmaniye Korkut Ata University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OsmaniyeKAU
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Sleep Quality
Keywords: sleep quality,; laughter yoga,; happiness,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control group (Experimental)
  Interventions: Other: yoga

INTERVENTIONS:
Other: yoga — laughter yoga

SUMMARY:
In this study, the effect of laughter yoga on sleep quality and happiness level in individuals with sleep problems will be investigated. Yoga exercises will be done for about 30 minutes with a laughter yoga instructor 3 days a week for a month.

ELIGIBILITY:
Inclusion Criteria:

individuals with sleep problems individuals without mental illness

Exclusion Criteria:

those who use sleeping pills those with mental disabilities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Laughter yoga improves sleep quality | 1-15. day
  The PSQI allows evaluating the quality and disturbances of sleep over one month. The questionnaire consists of 19 self-assessed questions that are categorized into 7 components: 1) sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disorders, 6) medication use to sleep, and 7) daytime sleepiness. Each component is classified in a score ranging from 0 to 3. The sum of the scores for these 7 components produces a score ranging from 0 to 21. It presents a cutoff point where it considers good sleep quality if PSQI≤5 and poor sleep quality if PSQI>5 21
Laughter yoga improves happiness | 1-15. day
  "Oxford Happiness Scale Short Form OHS-F", developed by Hills and Argyle (2002) and adapted into Turkish by Dogan and Cotok (2011) was used. Oxford Happiness Scale consists of 7 expressions in one sub-dimension. The expressions on the 5-item Likert scale are answered as (1) Disagree - (5) Completely agree.
Laughter yoga improves sleep quality | 30. DAY
  The PSQI allows evaluating the quality and disturbances of sleep over one month. The questionnaire consists of 19 self-assessed questions that are categorized into 7 components: 1) sleep quality, 2) sleep latency, 3) sleep duration, 4) sleep efficiency, 5) sleep disorders, 6) medication use to sleep, and 7) daytime sleepiness. Each component is classified in a score ranging from 0 to 3. The sum of the scores for these 7 components produces a score ranging from 0 to 21. It presents a cutoff point where it considers good sleep quality if PSQI≤5 and poor sleep quality if PSQI>5 21
Laughter yoga improves happiness | 30. day
  "Oxford Happiness Scale Short Form OHS-F", developed by Hills and Argyle (2002) and adapted into Turkish by Dogan and Cotok (2011) was used. Oxford Happiness Scale consists of 7 expressions in one sub-dimension. The expressions on the 5-item Likert scale are answered as (1) Disagree - (5) Completely agree.

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Sevgi ÜNAL ASLAN, Principal Investigator — OSMANİYE KORKUT ATA UNİVERSİTY
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No